CLINICAL TRIAL: NCT02498990
Title: Long-term Metabol Control After Weight Reduction With Low Calorie Diet in Type 2 Diabetes
Brief Title: Low Calorie Diet and Diabetes
Acronym: LCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Johan Hoffstedt, Associate Professor, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/628-31
Record Dates: First submitted 2015-07-03; First posted 2015-07-15 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus Type 2; Dyslipidemia; Non-alcoholic Fatty Liver Disease; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias; Non-alcoholic Fatty Liver Disease; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Weight reduction (Experimental)
  Interventions: Behavioral: Low calorie diet followed by life style intervention

INTERVENTIONS:
Behavioral: Low calorie diet followed by life style intervention — 1. Low calorie diet of 800 kcal/day for 7 weeks.
  2. Life style intervention for the remaining study period

SUMMARY:
The primary hypothesis is to investigate whether a low calorie diet for 7 weeks followed by continuous lifestyle advice is an effective option to achieve an improvement in glucose control as measured by HbA1c after 52 and 104 weeks as compared to baseline values in obese type 2 diabetes patients on either tablet or insulin treatment. The secondary hypothesis is to investigate whether the weight reduction therapy also has significant impact on various anthropometric, clinical and metabolic parameters associated with obesity.

DETAILED DESCRIPTION:
This is a prospective study on the impact of low calorie diet followed by a weight maintenance program on 12 and 24 month glucose control in a cohort of patients with obesity and diabetes mellitus. The study will consist of 3 phases:

1. Screening period (up to 12 weeks).
2. Low calorie diet weeks 1-9. Seven weeks of low-calorie diet including 800 kcal/day followed by 2 weeks of gradual introduction of normal diet of eventually 1500-2000 kcal/day, i.e. 600 kcal/day deficit, based on present body weight and sex. At entry of the LCD-period, all medication for diabetes mellitus, with the exception of metformin and insulin, will be removed. During the LCD-period, insulin treatment will gradually be reduced and, if possible, withdrawn. Patients will perform daily self-monitoring of fasting and post-prandial plasma glucose. At each visit, which will take place once a week, the patients will see a physician, a nurse and a dietician. The patients will be given specific advice to increase their physical activity. Patients will remain on medication for dyslipidemia. Blood pressure will be measured at each visit and in case of blood pressure < 110/70 mmHg and/or in case of symptoms associated with hypotension including dizziness, medication for hypertension will be reduced or removed.
3. Weight-maintenance program weeks 10-52.
4. Follow up visits at months 15, 18, 21 and 24.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women of age 18-65 years at screening.
2. Diagnosis of type 2 diabetes mellitus.
3. BMI > 30 kg/m2.
4. HbA1c > 52 mmol/mol.
5. Stable weight ± 5% for at least 12 weeks prior to screening.
6. Informed consent must be obtained by each subject before enrollment in the study.

Exclusion Criteria:

1. Pregnant or brest-feeding women or women who are planning to become pregnant or breast-feeding.
2. Type 1 diabetes mellitus or secondary forms of diabetes including pancreatic injury, cushing syndrome etc.
3. Clinically significant diabetic complications
4. Clinically symptomatic gastrointestinal or hepatic disease.
5. History of gastric bypass, antrectomy or small bowel disease.
6. History of pancreatitis.
7. Myocardial infarction within the past six months.
8. Symptomatic ischemic heart disease, heart failure or stroke.
9. Atrial fibrillation.
10. Patients on treatment with warfarin.
11. Diagnosed and/or treated malignancy within the past 5 years.
12. Any of the following laboratory abnormalities at screening:

    * ALT and/or AST > 3 times the upper limit of the normal range.
    * Serum creatinine levels > 130 µmol/l.
    * Clinically significant TSH out of the normal range.
    * Uric acid > 50% above normal level.
13. History of alcohol or other substance abuse within the past 2 years.
14. Psychiatric disease including eating disorder, bulimia nervosa, depression, anxiety, psychotic disease.
15. Potentially unreliable patients and those judged by the investigator to be unsuitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-08; Primary Completion 2024-02 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in HbA1c (mmol/mol) at 12 and 24 months | 12 months and 24 months

SECONDARY OUTCOMES:
Change from Baseline in BMI (kg/m2) at 7 weeks, 6,12, and 24 months | 7 weeks, 6, 12 and 24 months
Change from Baseline in Liver Fat (Controlled Attenuation Parameter, db/m) at 7 weeks, 6, 12 and 24 months | 7 weeks, 6, 12 and 24 months
  Liver Fat Measured by Fibroscan
Change from Baseline in Cholesterol (mmo/l) and Triglycerides (mmol/l) at 7 weeks, 6, 12 and 24 months | 7 weeks, 6,12 and 24 months
Change from Baseline in 2-hour Glucose (mmol/l) and Insulin (mU/l) by Glucose tolerance test at 7 weeks, 6, 12 and 24 months | 7 weeks, 6,12, 24 months
  Glucose tolerance test: oral administration of 75 g Glucose

CONTACTS AND LOCATIONS:
Overall Officials: Johan Hoffstedt, MD, PhD, Principal Investigator — Karilonska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden